CLINICAL TRIAL: NCT00589823
Title: A Multicentre, Double-Blind, Double-Dummy, Two-Phase Crossover Study of Fentanyl Citrate Nasal Spray Compared to Immediate Release Morphine Sulphate in the Treatment of BTCP in Subjects Taking Regular Opioid Therapy
Brief Title: Efficacy and Safety Study of Nasalfent for Treatment of Breakthrough Cancer Pain in Patients Taking Regular Opioids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Archimedes Development Ltd (Industry)
Responsible Party: Mark Watling, Group Medical Director, Archimedes Development Ltd
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CPO44/06/FCNS
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Cancers, Pain
Keywords: Pain; Cancer; Breakthrough
MeSH Terms: conditions — Neoplasms; Pain | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Immediate Release Morphine sulphate capsules taken at start of relevant BTCP episode. Each episode treated with either this medication OR the experimental comparator.
  Interventions: Drug: Fentanyl citrate
- 2 (Experimental): Nasalfent spray taken at start of relevant BTCP episode. Each episode to be treated with either this medication OR the active comparator (IRMS)
  Interventions: Drug: Immediate release morphine sulphate

INTERVENTIONS:
Drug: Fentanyl citrate — nasal spray, 100, 200, 400 or 800 mcg dosage according to need, to treat up to four episodes of BTCP per day
  Other Names: FCNS; Nasalfent
  Arms: 1
Drug: Immediate release morphine sulphate — drug dose as required by patient taken to treat up to four epsiodes of BTCP per day
  Other Names: IRMS
  Arms: 2

SUMMARY:
Cancer patients taking regular medication for their pain often still have episodes of severe pain that 'break through' despite their background pain treatment. Fentanyl is a strong, short-acting painkiller often used to treat this 'breakthrough' pain. Nasalfent contains fentanyl in a patented drug delivery system called PecSys and is given via a simple nasal spray. This study will test the efficacy and safety of Nasalfent compared to Immediate Release Morphine Sulphate in the treatment of breakthrough cancer pain.

DETAILED DESCRIPTION:
Current treatments for breakthrough cancer pain (BTCP)work too slowly to meet the fast onset of most BTCP episodes, they continue to act longer than the episode of pain lasts and so can have unwanted side effects due to this 'over treatment' of the pain episode. In addition many cancer patients have oral problems which make taking pain relief medication by mouth uncomfortable for the patient. Nasalfent is administered via the nose as a simple spray and can be taken by patients or given by their carers. The nasal route is a common way to administer medication for example in the treatment of migraine or allergy. At any time during the study the patient may take their regular treatment for BTCP should they so wish.

This study will compare the time of onset and degree of pain relief of Nasalfent to that of Immediate Release Morphine Sulphate. The safety of the two treatment options will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give consent
* Women of childbearing potential must have a) negative urine pregnancy test b) not be breast feeding c) agree to practice a reliable form of contraception
* Diagnosis of cancer
* Taking at least 60mg oral morphine or equivalent as 24 hour treatment for cancer-related pain
* Experiencing on average 1 - 4 episodes of breakthrough cancer pain per day usually controlled by rescue pain medication
* Able (or via caregiver) to evaluate and record pain relief, assess medication performance at set times after dosing, record adverse events, record each use of the study drug or rescue medication in a diary
* Able to be up and about for 50% of the day or greater

Exclusion Criteria:

* Intolerance to opioids or fentanyl
* rapidly increasing/uncontrolled pain
* pain that is not cancer-related

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pain Relief | Various time points

SECONDARY OUTCOMES:
Pain Relief at various time points | Various time points

CONTACTS AND LOCATIONS:
Overall Officials: Marie Fallon, Principal Investigator — Western General Hospital, Edinburgh Cancer Centre
Locations (1):
- Prof Fallon, Edinburgh, United Kingdom